CLINICAL TRIAL: NCT03252548
Title: Clinical Characteristics and Prognosis of Primary Immunodeficiency Disease (PID) in Chinese Children
Brief Title: Pediatric Primary Immunodeficiency Disease (PID) in China
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Beijing Children's Hospital (Other)
Collaborators: Capital Institute of Pediatrics, China (Other); Shenzhen Children's Hospital (Other Government)
Responsible Party: Principal Investigator, Kunling Shen, Chief of China National Clinical Research Center for Respiratory Diseases, Beijing Children's Hospital
Other Study IDs: BCHlung006
Record Dates: First submitted 2017-08-15; First posted 2017-08-17 (Actual); Last update posted 2018-01-03 (Actual); Status verified 2017-05

CONDITIONS: Primary Immunodeficiency Disease
MeSH Terms: conditions — Primary Immunodeficiency Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a prospective cohort study of children diagnosed with primary immunodeficiency disease (PID). The aim is to investigate the clinical characteristics and prognosis of PID in Chinese children.

DETAILED DESCRIPTION:
Primary immunodeficiency disease (PID) is a group of rare and fatal disease. However, the research about clinical characteristics, treatment, management and prognosis of Chinese children with PID is still not perfect and there is no basic and large database. Therefore, this study is conducted, in order to set up a complete database and long term follow up of Chinese children with PID, and establish foundations for basic research and precise medicine.

This study is divided into two parts. In part one, pediatric patients with PID in the past 10 years will be collected retrospectively by review medical records from these centers, and investigate the clinical features and prognosis. In part two, all new cases with suspected PID will be collected. Clinical symptoms, physical examination, blood tests, and humoral and cellular immune functions will be detected. Gene tests would be done when necessary to confirm the diagnosis. Then follow up at 6-moth, 1-year, 2-year, 3-year, 4-year and 5-year respectively. The trial will be completed in 60 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age: from neonates to 18 years old
2. Fulfilling the one of the followings:

   1. Severe infection after vaccination (BCG, polio arthritis pill)
   2. Chronic/recurrent ear infection, sinus infections and respiratory tract infection
   3. Recurrent, deep skin or deep-seated infections
   4. Boys with early period and refractory thrombocytopenia
   5. Infants with obviously decreased absolute number of lymphocytes
   6. Severe allergy with infection
   7. Infant diabetes with severe diarrhea
   8. Boys with severe Epstein-Barr virus infection
   9. Infants with hepatosplenomegaly and generalized lymphadenopathy
   10. Infantile hemophagocytic syndrome
   11. Failure of an infant to gain weight or grow normally
   12. Persistent thrush in mouth or fungalinfection on skin
   13. Family history of primary immunodeficiency
   14. Invasive pneumococcal infection
   15. Erythrodermic psoriasis
3. Gene test confirmed PID pediatric patients

Exclusion Criteria:

Subject will be excluded if she or he would not enroll into this study

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children who was confirmed diagnosis as PID at the certain hospitals
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Frequencies of severe infection of children with PID | 60 months
  Times of severe infection attack will be recorded every year from baseline to 60 months, assessed by questionnaire

SECONDARY OUTCOMES:
Life quality of children with PID | 60 months
  Life Quality Questionnaire, once for every year
Complications of children with PID | 60 months
Long-term changes on lung function of children with PID | 60 months

CONTACTS AND LOCATIONS:
Overall Officials: kunling shen, MD,PhD, Study Director — Beijing Children's Hospital, Capital Medical University, China; jianxin he, MD,PhD, Principal Investigator — Beijing Children's Hospital, Capital Medical University, China

IPD SHARING:
Plan to Share IPD: No